CLINICAL TRIAL: NCT05993338
Title: Assessment of Pulmonary Artery Pressure in COVID-19 Survivors Using Right Heart Catheterization
Brief Title: Pulmonary Artery Pressure in COVID-19 Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University Hospital (Other)
Responsible Party: Principal Investigator, Mohamed Abd Elmoniem Mohamed, Assistant lecturer chest medicine-Mansoura univerisity-Mansoura-Egypt, Mansoura University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: MD.22.04.638
Record Dates: First submitted 2023-08-13; First posted 2023-08-15 (Actual); Last update posted 2024-06-17 (Actual); Status verified 2024-06

CONDITIONS: Pulmonary Hypertension Secondary
Keywords: pulmonary artery pressure; COVID-19 survivors; right heart catheterization

STUDY DESIGN:
Intervention Model Description: assess pulmonary hemodynamics in COVID-19 survivors
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- assess pulmonary hemodynamics in COVID-19 survivors (Experimental): COVID-19 survivors from a moderate/severe COVID-19 pulmonary infection according to WHO COVID-19 clinical severity classification, ≥ 18 years, with residual symptoms and signs suggestive of pulmonary hypertension and not explained by other condition
  Interventions: Diagnostic Test: right heart catheterization (RHC).

INTERVENTIONS:
Diagnostic Test: right heart catheterization (RHC). — Assessment of pulmonary artery pressure in COVID-19 survivors using right heart catheterization (RHC).

SUMMARY:
Post COVID-19 pulmonary hypertension can develop as a result of lung parenchymal damage and altered pulmonary circulation induced by COVID-19 infection. It has been proposed that this type of PH should be considered a combination between PH of group 3 (due to interstitial fibrosis and alveolar inflammation) and 4 (induced by thrombotic/thromboembolic processes, endothelial injury, or, at least, hypoxic vasoconstriction). Right heart catheterization (RHC) is the gold standard for assessing pulmonary hemodynamics and is mandatory for confirming the diagnosis of pulmonary hypertension (PH), assessing the severity of hemodynamic impairment, and performing vasoreactivity testing in selected patients

DETAILED DESCRIPTION:
Coronavirus disease 2019 (COVID-19), the highly contagious viral illness caused by severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2), has had a catastrophic effect on the world's demographics resulting in more than 3.8 million deaths worldwide, emerging as the most consequential global health crisis since the era of the influenza pandemic of 1918. COVID-19 survivors may experience persistent symptoms affecting different organ systems after the acute phase of infection. Early reports suggest residual effects of SARS-CoV-2 infection, involving respiratory, cardiovascular, musculoskeletal, integumentary, gastrointestinal, endocrine, and neurological systems. Post-acute COVID-19 could be defined as persistent symptoms and/or delayed or long-term complications of SARS-CoV-2 infection beyond 4 weeks from the onset of symptoms. It is further divided into two categories: (1) subacute or ongoing symptomatic COVID-19, which includes symptoms and abnormalities present from 4-12 weeks beyond acute COVID-19; and (2) chronic or post-COVID- 19 syndrome, which includes symptoms and abnormalities persisting or present beyond 12 weeks of the onset of acute COVID-19 and not attributable to alternative diagnoses. Pulmonary hypertension (PH) is a clinical disorder involving multiple pathophysiological processes that ultimately affect the vasculature within the lungs.

According to the 6th World Symposium on Pulmonary Hypertension, pulmonary hypertension (PH) is defined by mean pulmonary arterial pressure (mPAP) >20 mmHg. "Pre-capillary PH" is considered if additionally pulmonary arterial wedge pressure (PAWP) is ≤15 mmHg and pulmonary vascular resistance (PVR) is ≥3 Wood units (WU). "Post-capillary PH" is defined as mPAP >20 mmHg with PAWP >15 mmHg. In the case of PVR <3 WU, we talk about "isolated post-capillary PH", while in the case of PVR ≥3 WU the criteria for "combined pre- and post-capillary PH" are fulfilled. Post COVID-19 pulmonary hypertension can develop as a result of lung parenchymal damage and altered pulmonary circulation induced by COVID-19 infection. It has been proposed that this type of PH should be considered a combination between PH of group 3 (due to interstitial fibrosis and alveolar inflammation) and 4 (induced by thrombotic/thromboembolic processes, endothelial injury, or, at least, hypoxic vasoconstriction). Right heart catheterization (RHC) is the gold standard for assessing pulmonary hemodynamics and is mandatory for confirming the diagnosis of pulmonary hypertension (PH), assessing the severity of hemodynamic impairment, and performing vasoreactivity testing in selected patients.

Hypothesis and assumptions:

We hypothesize that pulmonary hypertension explain some of residual symptoms in COVID-19 survivors.

Aim of work:

The aim of this study is to assess pulmonary hemodynamics in COVID-19 survivors.

ELIGIBILITY:
Inclusion Criteria:

* COVID-19 survivors from a moderate/severe COVID-19 pulmonary infection according to WHO COVID-19 clinical severity classification , ≥ 18 years, with residual symptoms and signs suggestive of pulmonary hypertension and not explained by other condition.

Exclusion Criteria:

* Previous diseases that could explain the existence of PH e.g. cardiovascular, pulmonary diseases or history of pulmonary thromboembolism.
* Hemodynamic instability.
* Absolute contraindications to RHC placement include:
* Infection at the insertion site.
* The presence of a right ventricular assist device.
* Insertion during cardiopulmonary bypass.
* Lack of consent.
* Relative contraindications to RHC placement include:
* Coagulopathy (INR >1.5), thrombocytopenia (platelet count <50,000/microL).
* Electrolyte disturbances.
* Severe acid-base disturbances.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2023-04-01 (Actual); Study Completion 2024-03-01 (Actual)

PRIMARY OUTCOMES:
Assessment of pulmonary artery pressure in COVID-19 survivors using right heart catheterization (RHC) | 1.5 year
  The pulmonary artery blood sample is withdrawn using the distal yellow port, and mixed venous oxygen saturation (SvO2) is obtained. Arterial saturation (SaO2) has to be obtained separately so as to determine the cardiac output (CO), using the Fick's method; CO, L/min = VO2/ [(SaO2 - SvO2) x Hb x 13.4)], where VO2 = 125 mL O2/min x BSA, In elderly patients (age ≥70 years), use 110 mL O2 x BSA for VO2, BSA = [(Height, cm x Weight, kg)/ 3,600]

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Abd Elmoniem, Study Director — assistant lecturer chest medicine Mansoura university
Locations (1):
- faculty of medicine Mansoura university, Al Mansurah, Egypt

IPD SHARING:
Plan to Share IPD: No